CLINICAL TRIAL: NCT06545734
Title: Effectiveness and Biological Mechanism of Direct Ischemic Post-conditioning for Acute Stroke Patients Due to Large Vessel Occlusion: A Randomized Controlled Pilot Trial
Brief Title: Effectiveness and Biological Mechanism of Direct Ischemic Post-conditioning for Acute Stroke Patients Due to Large Vessel Occlusion
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Huanhu Hospital (Other)
Responsible Party: Principal Investigator, Ming Wei, Chief Physician, Tianjin Huanhu Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJHH-2024-WM28
Record Dates: First submitted 2024-08-01; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Stroke, Acute; Neuroprotection; Ischemic Conditioning
Keywords: Stroke, Acute; Large Vessel Occlusion; Neuroprotection
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endovascular therapy (Active Comparator)
  Interventions: Procedure: Endovascular therapy
- Endovascular therapy plus direct ischemic post-conditioning (Experimental)
  Interventions: Procedure: Direct Ischemic Post-conditioning; Procedure: Endovascular therapy

INTERVENTIONS:
Procedure: Direct Ischemic Post-conditioning — After thrombectomy, the balloon was inflated to a pressure of no more than 4 atm at the occlusion site to block blood flow for 2 minutes, as confirmed by angiography. The balloon was then deflated, allowing blood flow to resume for 2 minutes. These steps were repeated four times.
  Arms: Endovascular therapy plus direct ischemic post-conditioning
Procedure: Endovascular therapy — Thrombectomy alone.

SUMMARY:
The goal of this clinical trial is to determine if direct ischemic post-conditioning (IPostC) can alleviate ischemic-reperfusion injury (I/R) in patients who have undergone endovascular thrombectomy (EVT). Additionally, the study aims to explore the underlying mechanisms of direct IPostC.

The primary questions this trial seeks to answer are:

1. Is direct IPostC effective for acute stroke patients with large vessel occlusion?
2. What are the underlying mechanisms of direct IPostC?

Participants will be randomly assigned to one of two groups: an EVT alone group or an EVT plus direct IPostC group. Direct IPostC will be administered immediately after EVT through four cycles of mechanical interruptions of reperfusion. We will evaluate outcomes based on final infarct volume, infarct volume growth, clinical parameters, and I/R-related imaging and laboratory biomarkers. Additionally, an exploratory multi-omics analysis will be conducted to uncover the detailed mechanisms of direct IPostC.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic stroke confirmed by CT or MRI.
2. Large vessel occlusion confirmed by CTA or MRA, including the intracranial internal 3. carotid artery (ICA) and middle cerebral artery (MCA M1/M2).

4. Recanalization of the occluded vessel at eTICI grade 2b/3, confirmed by DSA after thrombectomy.

5. The patient or legally authorized representative has signed an informed consent form.

Exclusion Criteria:

1. Inability to perform an MRI or CT scan for any reason.
2. Presence of any condition that would interfere with neurological assessment or any psychiatric disorders.
3. Stroke onset accompanied by seizures, resulting in the inability to obtain an accurate NIHSS baseline.
4. Pregnancy.
5. Presence of other serious, advanced, or terminal illnesses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-05 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Final Infarct volume | 24(-6/+12) hours after procedure
  Infarct volume at 24 (-6/+12) hours postoperatively
Infarct Volume Growth | 24(-6/+12) hours after procedure
  Infarct volume at 24 (-6/+12) hours - Infarct volume at baseline; Infarct volume at 24 (-6/+12) hours - Infarct volume at 2 hours

SECONDARY OUTCOMES:
Change in NIHSS between baseline and 2 hours | 2 hours after procedure
  NIHSS at 2 hours - NIHSS at baseline
Change in NIHSS between baseline and 24 hours | 24 hours after procedure
  NIHSS at 24 hours - NIHSS at baseline
Functional Independence at 90 days | 90 days after randomization
  The proportion of mRS 0-2 at 90 days
Functional Independence at 5 days or discharge | 5 days or at discharge after randomization
  The proportion of mRS 0-2 at 5 days or discharge
Blood brain barrier permeability at 72 hours | 72 hours after procedure
  This is quantified by ktrans value through MR

OTHER OUTCOMES:
Difference in Peripheral circulating immune cells counts | 1, 3 and 5 days after procedure
  Immune cell counts acquired from CBC.
Difference in lymphocyte phenotyping | PBMC isolated from peripheral venous blood at 24 hours
  CD4 T cells, CD8 T cells, B cells, NK cells count by flow cytometry.
Difference in expression of genes associated with T cell polarization | PBMC isolated from peripheral venous blood at 24 hours
  TBX21, GATA3, RORC and FOXP3
Difference in cytokines and chemokines associated with T cell polarization and recruitment | Serum isolated from peripheral venous blood at 24 hours
  IL-1β, IL-18, IL-17, IL-10, IFN-γ, TNF-α, IL-6, CX3CL1, CXCL10, CCL17

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes